CLINICAL TRIAL: NCT04975269
Title: Double-blind Randomized Acetazolamide Trial in Normal Pressure Hydrocephalus
Brief Title: Acetazolamide Trial in Normal Pressure Hydrocephalus
Acronym: DRAIN
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Collaborators: Uppsala University (Other); Swedish Society for Medical Research (Other)
Responsible Party: Principal Investigator, Johan Virhammar, Principal investigator, Uppsala University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NPH-01
Record Dates: First submitted 2021-06-15; First posted 2021-07-23 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Idiopathic Normal Pressure Hydrocephalus (INPH)
Keywords: normal pressure hydrocephalus; iNPH; Acetazolamide; Diamox; RCT
MeSH Terms: conditions — Hydrocephalus, Normal Pressure | interventions — Acetazolamide

STUDY DESIGN:
Intervention Model Description: Double-blind randomized trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acetazolamide (Active Comparator): Acetazolamide (active)
  Interventions: Drug: Acetazolamide
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetazolamide — Target dose: 500 mg / day
  Other Names: Diamox
  Arms: Acetazolamide
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A pharmacological treatment to patients with normal pressure hydrocephalus (NPH) is missing. The aim is to investigate if acetazolamide given to patients with NPH improves gait function and study the pathophysiological mechanisms leading to reduced symptoms.

Patients will be randomized to acetazolamide or placebo and duration of treatment will be from diagnosis to the day of shunt surgery. Target dose is 500 mg/day. Study design is a double-blind randomized controlled trial and the plan is to include 42-50 patients. The study is investigator-initiated without financial sponsorship from the industry.

DETAILED DESCRIPTION:
Background: The only available treatment for normal pressure hydrocephalus (NPH) is implantation of a neurosurgical shunt system that reduces symptoms in two out of three cases. Postoperative complications are common, causing reoperations in 20-30% within the first years after surgery. A pharmacological treatment is missing.

In three previous studies, acetazolamide, a reversible inhibitor of the carbonic anhydrase enzyme, was used as treatment off-label. In the first of these studies, 15 patients with NPH were treated with doses 250-500 mg/day and 10 patients improved (Aimard G et. al.). The second study was a case report of one patient with NPH who improved after receiving the dose 500 mg/day (Garcia-Gasco P et. al.). The most recent study used doses of 125-375 mg/day and included 8 patients of whom 5 improved. Furthermore, the last study reported a reduction of the periventricular edema that is often present in the white matter close to the lateral ventricles in patients with NPH (Alperin N et. al.). These three studies were open label with no blinding or control group.

Study design: Study design is a double-blind randomized placebo-controlled trial. The study is investigator-initiated without financial sponsorship from the industry. The plan is to consecutively include 42-50 patients with NPH. Patients will be randomized to acetazolamide or placebo and take the study drug from diagnosis (baseline) to admission for shunt surgery. Waiting time for shunt surgery at the center of the study is approximately 4-8 months at the moment. The dose will be titrated to 250 mg x 2 during 4-6 weeks. Two phone visits with a study nurse and routine blood samples are controlled during the titration phase to rule out side effects.

Evaluations of clinical symptoms and blood samples for blood biomarkers are collected at baseline, after 3 months and when the study drug is stopped. Lumbar cerebrospinal fluid (CSF) is collected at baseline and intraventricular CSF is collected during shunt surgery. All patients are investigated after shunt surgery, 3 months postoperatively with evaluation of symptoms and blood samples. Blood- and CSF samples are stored in a biobank.

In a subgroup of 24-26 patients, an MRI of the brain is performed before the start of study drug and after 3 months. In this subgroup also assessments of symptoms and blood samples for analysis of plasma biomarkers will be collected in connection with the MRI scans.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of idiopathic normal pressure hydrocephalus according to international guidelines
2. Age ≥ 50 years and ≤ 82 years
3. Cognitive function with Mini-Mental State Examination > 20 points or cognitive domain of iNPH scale ≥ 30 points.
4. MRI image characteristic of normal pressure hydrocephalus, defined as callosal angle < 90 degrees and dilated lateral ventricles or pattern of disproportionately enlarged subarachnoid space hydrocephalus (DESH).
5. Signed informed consent form

Exclusion Criteria:

1. Exclusion criteria for MRI examination
2. Participation in another medical trial
3. Other disease likely to impact the symptoms of the patient
4. Wheelchair user or unable to walk without support
5. Reduced kidney function with GFR < 50
6. Reduced liver function (increased INR or alanine transaminase concentrations in plasma elevated more than 1.5 times reference values)
7. Known heart failure
8. Low concentrations of electrolytes in blood plasma that, according to the investigator, prevents participation in the study
9. Angle-closure glaucoma
10. Allergy to acetazolamide, sulfonamides, or sulfonamide derivatives
11. Treatment with phenytoin, valproate, carbamazepine, lithium, oral anticoagulants, thiazide-diuretics, or acetylsalicylic acid > 100 mg/day
12. Inability to swallow capsules of the same size as the investigational medicinal products (will be tested using empty capsules when the patient is asked to participate in the study)
13. Average walking time for the three walking tests < 10.5 seconds for men and < 11.5 seconds for women.
14. Average walking time for the three walking tests > 50 seconds
15. Inability to comply with the study treatment independently, and a concurrent lack of individuals to help the patient comply with the treatment during the study period
16. Fertile woman without highly effective contraception. A Fertile woman will be tested with pregnancy test before inclusion is possible.

Ages: 50 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportional change in gait function | Change from baseline gait function immediately after intervention (at time of shunt surgery)
  Gait function is determined by one variable that is calculated as the mean time and number of steps of three different gait tests: 10 meter walking in self chosen speed, timed up and go test (TUG) and 3 m walking backwards.
  The two fastest attempts of three attempts for each test are documented. The mean time and number of steps of the two fastest attempts for the three tests are calculated to a single variable and the proportional difference between study visits is used as the primary outcome variable.

SECONDARY OUTCOMES:
Change in idiopathic normal pressure hydrocephalus (iNPH) scale | Change from baseline iNPH-scale score immediately after intervention (at time of shunt surgery)
  Swedish idiopathic normal pressure hydrocephalus (iNPH) scale that is a combination of subscales for gait, balance, cognition and continence. Minimum value is 0 and maximum value is 100. High values indicate better function.
Change in volume of periventricular hyperintensities | Change from baseline at 3 months
  Measured using volumetric MRI
Change in cerebral blood perfusion | Change from baseline at 3 months
  Measured using pseudo continuous arterial spin labeling (MRI perfusion)
Change in quantified CSF flow in cerebral aqueduct | Change from baseline at 3 months
  Measured using phase contrast MRI
Change in parenchymal water content | Change from baseline at 3 months
  Measured using Synthetic MRI
Change in cerebral myelin volume | Change from baseline at 3 months
  Measured using Synthetic MRI
Changes in plasma biomarkers | Change from baseline immediately after intervention (at time of shunt surgery)
  Change in plasma levels of neurofilament light chain protein, Total-tau, amyloid beta-42, glial fibrillary acidic protein will be measured using Quanterix (SIMOA).
Change in CSF biomarkers | Change from baseline immediately after intervention (at time of shunt surgery)
  CSF levels of neurofilament light chain protein, Total-tau, amyloid beta-42, glial fibrillary acidic protein will be measured using Quanterix (SIMOA).
Changes in plasma and CSF proteins | Change from baseline immediately after intervention (at time of shunt surgery)
  Semi-quantified levels of approximately 200 proteins are measured with proximity extension assay (Neurology panel and Neuro exploratory panel, Olink.com).
Patients self reported assessment of symptoms | Change from baseline immediately after intervention (at time of shunt surgery)
  Gait, cognition, continence, balance, activities of daily life and quality of life is rated by patients on a questionnaire using 4-level scales.
Change in Euro-Quality of Life-5 dimension-5L (EQ-5D-5L) descriptive system | Change from baseline EQ-5D-5L score immediately after intervention (at time of shunt surgery)
  Measured using EQ-5D-5L using the descriptive system.
Change in Euro-Quality of Life-5 dimension-5L (EQ-5D-5L) VAS | Change from baseline EQ-5D-5L score immediately after intervention (at time of shunt surgery)
  Measured using the visual analogue scale (VAS) in EQ-5D-5L.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Virhammar, MD, PhD, Principal Investigator — Department of Neuroscience, Uppsala University
Locations (1):
- Department of Clinical Neurophysiology, Neurosurgery and Neurology, Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in any publications from this study, can be shared after deidentification.
Supporting Information: Study Protocol
Time Frame: From publication of the first article from this study, ending 10 years following the last published article from this study.
Access Criteria: Researchers who provide a methodologically sound proposal can contact the principal investigator of the study.

REFERENCES:
- [Background] Aimard G, Vighetto A, Gabet JY, Bret P, Henry E. [Acetazolamide: an alternative to shunting in normal pressure hydrocephalus? Preliminary results]. Rev Neurol (Paris). 1990;146(6-7):437-9. French. PMID 2399408
- [Background] Adams RD, Fisher CM, Hakim S, Ojemann RG, Sweet WH. SYMPTOMATIC OCCULT HYDROCEPHALUS WITH "NORMAL" CEREBROSPINAL-FLUID PRESSURE. A TREATABLE SYNDROME. N Engl J Med. 1965 Jul 15;273:117-26. doi: 10.1056/NEJM196507152730301. No abstract available. PMID 14303656
- [Background] Garcia-Gasco P, Salame Gamarra F, Tenllado Doblas P, Chazarra Talens C. [Complete resolution of chronic hydrocephalus of adult with acetazolamide]. Med Clin (Barc). 2005 Apr 9;124(13):516-7. doi: 10.1157/13073568. No abstract available. Spanish. PMID 15847775
- [Background] Alperin N, Oliu CJ, Bagci AM, Lee SH, Kovanlikaya I, Adams D, Katzen H, Ivkovic M, Heier L, Relkin N. Low-dose acetazolamide reverses periventricular white matter hyperintensities in iNPH. Neurology. 2014 Apr 15;82(15):1347-51. doi: 10.1212/WNL.0000000000000313. Epub 2014 Mar 14. PMID 24634454
- [Background] Relkin N, Marmarou A, Klinge P, Bergsneider M, Black PM. Diagnosing idiopathic normal-pressure hydrocephalus. Neurosurgery. 2005 Sep;57(3 Suppl):S4-16; discussion ii-v. doi: 10.1227/01.neu.0000168185.29659.c5. PMID 16160425
- [Background] Hellstrom P, Klinge P, Tans J, Wikkelso C. A new scale for assessment of severity and outcome in iNPH. Acta Neurol Scand. 2012 Oct;126(4):229-37. doi: 10.1111/j.1600-0404.2012.01677.x. Epub 2012 May 16. PMID 22587624